CLINICAL TRIAL: NCT01225510
Title: A Phase 2 Trial Of PF-04856884 (CVX-060), A Selective Angiopoietin-2 (Ang-2) Binding CovX-body, In Patients With Recurrent Glioblastoma
Brief Title: A Trial Of PF-04856884 In Patients With Recurrent Glioblastoma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B1131003
Record Dates: First submitted 2010-10-19; First posted 2010-10-21 (Estimated); Last update posted 2015-03-11 (Estimated); Status verified 2015-03

CONDITIONS: Glioblastoma
Keywords: recurrent glioblastoma multiforme (GBM); CVX-060; PF-04856884; phase 2; open-label; bevacizumab; anti-angiogenic
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Primary Cohort (Experimental)
  Interventions: Biological: PF-04856884
- Exploratory Cohort (Experimental)
  Interventions: Biological: PF-04856884

INTERVENTIONS:
Biological: PF-04856884 — PF-04856884 at a dose of 15 mg/kg/week
  Other Names: CVX-060
  Arms: Primary Cohort
Biological: PF-04856884 — PF-04856884 at a dose of 15 mg/kg/week
  Other Names: CVX-060
  Arms: Exploratory Cohort

SUMMARY:
Angiopoietin-2 (Ang-2) is a protein in the body which destabilizes blood vessels and is important in stimulating tumor blood vessels. There is evidence suggesting that Ang-2 may be important for the growth and progression of Glioblastoma multiforme (GBM). PF- 04856884 (CVX-060) is a compound which binds Ang-2 and prevents its activity. The hypothesis is that PF-04856884 will be safe and effective in patients with recurrent Glioblastoma multiforme (GBM).

DETAILED DESCRIPTION:
Notification of study being cancelled resulted in update in overall status change from "not yet recruiting" to "withdrawn."

ELIGIBILITY:
Inclusion Criteria:

* Tumor eligibility: Primary Cohort: Measurable disease; Exploratory Cohort: Measurable disease as defined above or non-measurable/evaluable disease (eg, progressing non-enhancing lesions).
* Histologically or cytologically confirmed recurrent GBM in 1st or 2nd relapse: Primary Cohort: Recurrence following radiation therapy and temozolomide, less than or equal to 2 prior chemotherapeutic regimens; Exploratory cohort: Prior radiation therapy, temozolomide, and bevacizumab, Recurrence of disease within 2-4 weeks of last bevacizumab dose.
* Stable dose of corticosteroids for greater than or equal to 5 days prior to baseline Magnetic Resonance Imaging (MRI)
* Adequate organ function
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Life expectancy greater than or equal to 12 weeks.

Exclusion Criteria:

* Patients who have previously received a trial drug containing the core platform antibody (eg, CVX-045, PF-04856884 (CVX-060), CVX-096, PF-05057459 (CVX-241), etc.).
* History of pathologic fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months of therapy.
* Evidence of bleeding diathesis or coagulopathy.
* Major surgical procedure (eg, craniotomy), open biopsy, significant traumatic injury within 28 days prior to therapy or anticipation of need for a major surgical procedure during the course of the trial.
* Minor surgical procedures, fine needle aspiration or core biopsies within 7 days prior to therapy.
* Serious non-healing wound, ulcer, or bone fracture.
* Active gastrointestinal bleeding, as evidenced by either hematemesis, hematochezia, or melena in prior 6 months.
* Hemoptysis >½ teaspoon per day within 1 week of enrollment.
* National Cancer Institute-Common Terminology Criteria for Adverse Events [NCI CTCAE] Grade 3 hemorrhage from any cause <4 weeks prior to enrollment.
* Participation in any investigational drug study within 28 days prior to study therapy.
* Evidence of preexisting uncontrolled hypertension
* Clinically significant cardiovascular disease within the 12 months prior to starting trial treatment
* Prolongation of the QT interval corrected [QTc] interval to >450 msec for men or >470 msec for women.
* History of allergic or anaphylactic reaction to any therapeutic or diagnostic monoclonal antibody or IgG-fusion protein.

Exclusion Criteria Specific for Primary Cohort

* Prior therapy with bevacizumab or other anti-Vascular Endothelial Growth Factor [VEGF] agents for the treatment of GBM.

Exclusion Criteria Specific for Exploratory Cohort

* Patients discontinued from prior bevacizumab or anti-VEGF agents due to toxicity.
* Patients who have failed 2 prior anti-VEGF therapies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-01; Primary Completion 2013-01 (Estimated); Study Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
Progression free survival rate at Month 6 (PFS6) defined as the patient progression free status at Month 6. | 1 year

SECONDARY OUTCOMES:
Corticosteroid doses at baseline and on-study | 4 months
Overall Response Rate (ORR) | 2 years
PFS defined as the time from 1st dose of study drug to the 1st documentation of disease progression or death from any cause, whichever comes first. | 2 years
Time to death is defined as the time from first study drug to death due to any cause. | 2 years
Overall survival (OS) defined as the time from first dose of study drug to death due to any cause. | 2 years
OS6 defined as the patient survival status at Month 6. The OS6 rate will be obtained as a Kaplan-Meier estimate of the time to death at Month 6. | 2 years
Immunogenicity determined by measuring anti-PF-04856884 antibodies following therapy | 4 months
Dynamic Contrast Enhanced Magnetic Resonance Imaging [DCE-MRI] endpoints to include changes from baseline volume transfer coefficient [Ktrans] and/or the initial area under the contrast agent concentration-time curve [IAUC] or Ki following therapy | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1131003&StudyName=A%20Trial%20Of%20PF-04856884%20In%20Patients%20With%20Recurrent%20Glioblastoma%20